CLINICAL TRIAL: NCT00245869
Title: Contrast-Enhanced Ultrasound and Neoadjuvant Chemotherapy of Breast Cancer: Relationship Between Early Vascular Changes of the Tumor and Late Tumoral Response
Brief Title: Ultrasound and Chemotherapy of Breast Cancer: Relationship Between Early Vascular Changes of the Tumor and Late Tumoral Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CT03-FD/COR
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2006-07

CONDITIONS: Breast Cancer
Keywords: Contrast-enhanced Ultrasound; Ultrasound Contrast agents, microbubbles; breast cancer; chemotherapy; vascularization
MeSH Terms: conditions — Breast Neoplasms; Neovascularization, Pathologic

INTERVENTIONS:
Procedure: Contrast-enhanced Ultrasound

SUMMARY:
This study intends to assess the ability of contrast-enhanced ultrasound to make the efficacy of chemotherapy in breast cancer precise.

This real-time noninvasive and feasible imaging technique allows us, the investigators at University Hospital Tours, to evaluate early vascular changes of breast tumors during treatment. These vascular changes may precede long-term tumoral regression. Imaging of primary breast lesions may be of value in the prediction of late treatment response.

An ultrasound will be performed before the initiation, and after the second and the last dose of chemotherapy.

To investigate the changes occurring in the vascularization of tumors, we will use an intravascular ultrasound contrast agent SonoVue (sulphur hexafluoride microbubbles).

This agent is a microbubbles preparation that is stable, resistant to pressure, and specifically designed to be used as a contrast agent for ultrasound imaging of angiogenesis.

DETAILED DESCRIPTION:
The main objective of the study is to evaluate the early vascular changes of the tumor during neoadjuvant chemotherapy compared to the clinical or MRI or histological response.

ELIGIBILITY:
Inclusion Criteria:

* Breast tumor (size equal to or greater than 3 cm.). Patients with diagnosis of benign breast tumor based on biopsy will be excluded from the study after the first ultrasound examination.
* Neoadjuvant chemotherapy is programmed when an epithelial carcinoma is diagnosed by histology.
* Performance status = 0, 1 or 2
* No previous surgery or local radiotherapy

Exclusion Criteria:

* Psychiatric disorders
* Vital threat due to other disease
* Vital prognosis < 3 months
* Biopsy of the lesion performed within 1 month before the ultrasonography
* Patient known to have a coronary syndrome
* Unstable angina and myocardial infarction
* Acute cardiac failure, Class III/IV cardiac failure
* Several arrhythmias
* Acute endocarditis
* Prosthetic valves

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-03; Study Completion 2007-02

PRIMARY OUTCOMES:
From contrast-enhanced ultrasound: Enhancement parameters derived from time-intensity curves

CONTACTS AND LOCATIONS:
Overall Officials: François Tranquart, PR, Study Director — Centre d'Innovation Technologique - CHRU Tours; Catherine LABBE, MD, Principal Investigator — CRLCC René Gauducheau 44805 ST HERBLAIN
Locations (1):
- University Hospital of Tours, Tours, France

REFERENCES:
- [Background] Singh S, Pradhan S, Shukla RC, Ansari MA, Kumar A. Color Doppler ultrasound as an objective assessment tool for chemotherapeutic response in advanced breast cancer. Breast Cancer. 2005;12(1):45-51. doi: 10.2325/jbcs.12.45. PMID 15657523
- [Background] Watermann D, Madjar H, Sauerbrei W, Hirt V, Prompeler H, Stickeler E. Assessment of breast cancer vascularisation by Doppler ultrasound as a prognostic factor of survival. Oncol Rep. 2004 Apr;11(4):905-10. PMID 15010893
- [Background] Folkman J. Angiogenesis in cancer, vascular, rheumatoid and other disease. Nat Med. 1995 Jan;1(1):27-31. doi: 10.1038/nm0195-27. PMID 7584949
- [Background] Hansen S, Grabau DA, Rose C, Bak M, Sorensen FB. Angiogenesis in breast cancer: a comparative study of the observer variability of methods for determining microvessel density. Lab Invest. 1998 Dec;78(12):1563-73. PMID 9881956
- [Background] Hansen S, Grabau DA, Sorensen FB, Bak M, Vach W, Rose C. The prognostic value of angiogenesis by Chalkley counting in a confirmatory study design on 836 breast cancer patients. Clin Cancer Res. 2000 Jan;6(1):139-46. PMID 10656442
- [Background] Smith IC, Welch AE, Hutcheon AW, Miller ID, Payne S, Chilcott F, Waikar S, Whitaker T, Ah-See AK, Eremin O, Heys SD, Gilbert FJ, Sharp PF. Positron emission tomography using [(18)F]-fluorodeoxy-D-glucose to predict the pathologic response of breast cancer to primary chemotherapy. J Clin Oncol. 2000 Apr;18(8):1676-88. doi: 10.1200/JCO.2000.18.8.1676. PMID 10764428
- [Background] Schelling M, Avril N, Nahrig J, Kuhn W, Romer W, Sattler D, Werner M, Dose J, Janicke F, Graeff H, Schwaiger M. Positron emission tomography using [(18)F]Fluorodeoxyglucose for monitoring primary chemotherapy in breast cancer. J Clin Oncol. 2000 Apr;18(8):1689-95. doi: 10.1200/JCO.2000.18.8.1689. PMID 10764429
- [Background] Denis F, Bougnoux P, Paon L, le Floch O, Tranquart F. Radiosensitivity of rat mammary tumors correlates with early vessel changes assessed by power Doppler sonography. J Ultrasound Med. 2003 Sep;22(9):921-9. doi: 10.7863/jum.2003.22.9.921. PMID 14510263
- [Background] Denis F, Colas S, Chami L, Louisot P, Le Floch O, Tranquart F, Bougnoux P. Changes in tumor vascularization after irradiation, anthracyclin, or antiangiogenic treatment in nitrosomethyl ureas-induced rat mammary tumors. Clin Cancer Res. 2003 Oct 1;9(12):4546-52. PMID 14555529
- [Background] Kook SH, Kwag HJ. Value of contrast-enhanced power Doppler sonography using a microbubble echo-enhancing agent in evaluation of small breast lesions. J Clin Ultrasound. 2003 Jun;31(5):227-38. doi: 10.1002/jcu.10172. PMID 12767017
- [Background] Solesvik OV, Rofstad EK, Brustad T. Vascular changes in a human malignant melanoma xenograft following single-dose irradiation. Radiat Res. 1984 Apr;98(1):115-28. PMID 6718687